CLINICAL TRIAL: NCT00338936
Title: A 52-week Extension to the Factorial Study to Evaluate the Efficacy and Safety of VAH631 (Valsartan and Hydrochlorothiazide Combined) and Alone in Essential Hypertensive Patients - Long Term Study of VAH631 in Patients With Essential Hypertension (Extension From B1303 Study) -
Brief Title: Long Term Study of VAH631 in Patients With Essential Hypertension (Extension From B1303 Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631B1303E1
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: Hypertension; Valsartan; Hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan + Hydrochlorothiazide

SUMMARY:
This study is designed to provide long-term safety and efficacy data for the combination doses of VAH (VAL/ HCTZ) 40/6.25mg and 80/12.5mg in essential hypertensive patients. The 350 patients (approximately) who have successfully finished the core trial CVAH631B1303 and signed consent for the extension will be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who successfully complete the core study (Protocol 1303)
* Outpatients

Exclusion Criteria:

* Presence of crucial protocol violation in Protocol 1303
* Patients who experienced any adverse events considered serious and drug related in Protocol 1303.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Assessment of safety through reporting of adverse events, serious adverse events and deaths over 52 weeks.

SECONDARY OUTCOMES:
Change from baseline in average sitting diastolic blood pressure after 52 weeks
Change from baseline in average sitting systolic blood pressure after 52 weeks
Change from baseline in average standing diastolic blood pressure after 52 weeks
Change from baseline in average standing systolic blood pressure after 52 weeks
Laboratory abnormalities after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma Ag, Study Director — Novartis Pharmaceuticals